CLINICAL TRIAL: NCT06177080
Title: Evaluation of the Active Phase of Delivery by Transperineal Ultrasound and the Place of Sonopartograph in Travay Follow-up in Term Pregnancy
Brief Title: Transperineal Ultrasound and the Place of Sonopartograph in Travay Follow-up in Term Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor Department of Obstetrics and Gynecology, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2011-KAEK-252021/10-13
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Intrapartum; Transperineal Ultrasound
Keywords: head symphysis distance; angle of progression; sonopartograph

STUDY DESIGN:
Intervention Model Description: 30 nulliparous and 70 multiparous total 100 singleton pregnant women measured descent angle and head symphysis distances by transperineal ultrasound in the active phase of labor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Definitions of active phase angle of progression, head symphysis distance and examination findings (Other): Definitions of active phase AOP and HSD and examination findings measured in each period according to the type of birth
  Interventions: Other: transperineal ultrasound

INTERVENTIONS:
Other: transperineal ultrasound — descent angle and head symphysis distances by transperineal ultrasound of active phase of labor women.

SUMMARY:
Investigators aimed to determine the progression of the descent angle and head symphysis distance measured by intrapartum transperineal ultrasound as an alternative to vaginal examination and bishop score, according to time and cervical dilatation and to draw a sonopartograph as a new indicator also aimed to evaluate the success of the use of transperineal ultrasound in the active phase of labor in predicting prolonged labor, duration and mode of of delivery.

DETAILED DESCRIPTION:
Descent angle and head symphysis distances by transperineal ultrasound of pregnant women who are in the active phase of labor was measured hourly in the first phase of the active phase (the period from 4 cm to full dilation of the cervical opening); every 15 minutes in the second phase of the active phase (time from full dilation to delivery of the baby) Cervical dilatation and head levels were noted by simultaneous digital vaginal examination. The physician who performed the imaging and the physician who made the vajinal examination worked independently of each other and did not see each other's results.

ELIGIBILITY:
Inclusion Criteria:

* multiparous pregnancy
* active phase in labor
* vertex position

Exclusion Criteria:

* multiple pregnancy
* BMI over 35
* preterm labor
* congenital anomalies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Transperineal ultrasound instead of digital vaginal examination | 7 months
  use of transperineal ultrasound in the active phase of labor in predicting prolonged labor, duration and mode of delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Nazlı YENIGUL, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No